CLINICAL TRIAL: NCT02183922
Title: Hypocaloric Diet With or Without Microencapsulated Fish Oil or Conjugated Linoleic Acid on Oxidative Stress and Cardiovascular Risk Factors in Women With Metabolic Syndrome Genotyped for Polymorphisms in the Genes PPAR Gamma 2 (Pro12Ala) and Adiponectin (G276T)
Brief Title: Microencapsulated Fish Oil or Conjugated Linoleic Acid in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Sofia Kimi Uehara, Doctor, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 181/10
Record Dates: First submitted 2014-06-27; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Insulin Resistance; Oxidative Stress; Lipid Profile; Blood Pressure; Anthropometric Measure
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- light fruit jam (Placebo Comparator): The placebo group received light fruit jam (15 g/day) during 12 weeks.
  Interventions: Dietary Supplement: light fruit jam
- microencapsulated fish oil (Experimental): The microencapsulated fish oil group received light fruit jam with microencapsulated fish oil (3 g/day) during 12 weeks.
  Interventions: Dietary Supplement: microencapsulated fish oil
- microencapsulated conjugated linoleic acid (Experimental): The microencapsulated conjugated linoleic acid group received light fruit jam with microencapsulated conjugated linoleic acid (3 g/day) during 12 weeks.
  Interventions: Dietary Supplement: microencapsulated conjugated linoleic acid

INTERVENTIONS:
Dietary Supplement: microencapsulated conjugated linoleic acid — The microencapsulated conjugated linoleic acid received light fruit jam with microencapsulated conjugated linoleic acid (3 g/day) during 12 weeks.
  Arms: microencapsulated conjugated linoleic acid
Dietary Supplement: microencapsulated fish oil — The microencapsulated fish oil group received light fruit jam with microencapsulated fish oil (3 g/day) during 12 weeks.
  Arms: microencapsulated fish oil
Dietary Supplement: light fruit jam — The placebo group received light fruit jam (15 g/day) during 12 weeks.
  Arms: light fruit jam

SUMMARY:
Our aim was to assess the effects of a hypocaloric diet, including diet fruit jelly with microencapsulated fish oil or conjugated linoleic acid or placebo, on anthropometry, body composition, insulin resistance and lipid profile in women with metabolic syndrome and genotype Pro12Pro in the PPAR gamma 2 gene.

ELIGIBILITY:
Inclusion Criteria:

* adults women (30-45 years old);
* diagnosis of metabolic syndrome, as defined by the International Diabetes Federation;
* Pro12Pro genotype in gene PPARγ2.

Exclusion Criteria:

Participants were excluded if they:

* Were allergic to strawberries or fish
* Were pregnant or lactating
* Took fatty acid supplements
* Had undergone bariatric surgery or were being treated nutritionally or pharmacologically for reducing BM, or had taken anti-obesity drugs during the previous three months

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2008-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Oxidative stress biomarker | Change from baseline at 12 weeks
  Plasma malondialdehyde levels

SECONDARY OUTCOMES:
Insulin resistance | Change from baseline at 12 weeks
  Homeostatic Model Assessment-Insulin Resistance index, adiponectin, glucose and insulin levels
Lipid profile | Change from baseline at 12 weeks
  Total cholesterol, LDL-cholesterol, VLDL-cholesterol, HDL-cholesterol and triglycerides serum levels and EPA, DHA and total conjugated linoleic acid plasma levels
Anthropometric measures | Change from baseline at 12 weeks
  Body weight, body mass index and waist circumference
Body composition measures | Change from baseline at 12 weeks
  Fat-free mass and fat mass
Blood pressure | Change from baseline at 12 weeks
  Systolic blood pressure and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Uehara, Nutritionist, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil